CLINICAL TRIAL: NCT00895726
Title: Open-Label, Pilot Phase I/II Study of the Efficacy and Safety of APD209 in Patients With Cachexia and Advanced Malignancy
Brief Title: Pilot Study of APD209 in Cancer Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC10004
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Cancer-related Cachexia
Keywords: cachexia; neoplasms
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APD209 (Experimental)
  Interventions: Drug: APD209

INTERVENTIONS:
Drug: APD209 — Oral tablets twice per day for 56 days

SUMMARY:
Primary Objective:

To assess the efficacy of APD209 in adult patients with active cachexia associated with advanced malignancy and not caused by simple starvation.

Secondary Objective:

To assess the safety of APD209 in patients with advanced malignancy and active cachexia.

ELIGIBILITY:
Inclusion Criteria:

* Involuntary loss of weight of >= 2% in 2 months or >= 5% in 6 months, and ongoing in recent weeks, without (or with successfully treated) secondary causes of impaired oral nutritional intake (simple starvation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Muscle size and function | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Fox, MB BChir, Study Director — Acacia Pharma Ltd
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, United Kingdom